CLINICAL TRIAL: NCT03673826
Title: Carfilzomib, Lenalidomide and Dexamethasone Versus Lenalidomide and Dexamethasone in High- Risk Smoldering Multiple Myeloma: A Randomized Phase II Study.
Brief Title: Carfilzomib, Lenalidomide and Dexamethasone Versus Lenalidomide and Dexamethasone in High- Risk SMM
Acronym: HO147SMM
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Stichting Hemato-Oncologie voor Volwassenen Nederland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HO147; 2017-000555-10 (EudraCT Number)
Record Dates: First submitted 2018-09-06; First posted 2018-09-17 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2023-10

CONDITIONS: Smouldering Myeloma
MeSH Terms: conditions — Smoldering Multiple Myeloma | interventions — carfilzomib; Dexamethasone; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A (Experimental): Rd combination (Cycles 1-9 lenalidomide 25 mg, dexamethasone 20 mg cycles 1-4 and 10 mg cycles 5-9); followed by extended lenalidomide dosing (10 mg days 1-21 of a 28 day cycle for 24 cycles).
  Interventions: Drug: Dexamethasone; Drug: Lenalidomide
- Arm B (Experimental): KRd combination (Cycles 1-9 carfilzomib 20/36 mg/m2, lenalidomide 25 mg, dexamethasone 20 mg cycles 1-4 and 10 mg cycles 5-9); followed by extended lenalidomide dosing (10 mg days 1-21 of a 28 day cycle for 24 cycles).
  Interventions: Drug: Carfilzomib; Drug: Dexamethasone; Drug: Lenalidomide

INTERVENTIONS:
Drug: Carfilzomib — 9 cycles 20/36mg/m2 days 1,2,8,9,15,16
  Arms: Arm B
Drug: Dexamethasone — 4 cycles 20 mg days 1,2,8,9,15,16,22,23 followed by 5 cycles 10mg days 1,2,8,9,15,16,22,23
Drug: Lenalidomide — 9 cycles 25mg days 1-21 followed by 24 extended dosing cycles 10mg days 1-21

SUMMARY:
Randomized (2:1) multi-center open-label phase II trial. Patients with high-risk SMM will be enrolled on the study and treated with KRd combination (Cycles 1-9 carfilzomib 20/36 mg/m2, lenalidomide 25 mg, dexamethasone 20 mg cycles 1-4 and 10 mg cycles 5-9) or Rd combination (Cycles 1-9 lenalidomide 25 mg, dexamethasone 20 mg cycles 1-4 and 10 mg cycles 5-9); followed by extended lenalidomide dosing (10 mg days 1-21 of a 28 day cycle for 24 cycles).

DETAILED DESCRIPTION:
Background of the study:

A recent study has shown that intervention with the use of novel agents in smoldering myeloma (SMM) resulted in prolonged PFS and OS without significant toxicity. A more recent pilot study in high-risk smoldering myeloma using carfilzomib, lenalidomide in combination with dexamethasone resulted in 100% CR rate and 10 out of 12 patients reached MRD negativity. These studies formed the rationale to compare the efficacy and safety of carfilzomib, lenalidomide and dexamethasone vs. lenalidomide, dexamethasone, both followed by 24 months of lenalidomide maintenance in high-risk SMM.

This study is designed to compare 2 treatment modalities to find the optimal treatment in efficacy and safety for highrisk SMM, to define new risk stratifiers for outcome to treatment in SMM and to better understand the biology of SMM.

Objective of the study:

The primary objective of the study is :

To assess the progression-free survival rate of KRd versus Rd in patients with high-risk SMM

Secondary objectives:

* To assess MRD status after 4 and 9 cycles induction treatment
* To assess the correlation between PFS and MRD
* To determine progression-free survival-2 (PFS2 )
* To determine duration of response (DOR)
* To determine overall survival (OS)
* To assess correlation of MRD status with PFS2, DOR and OS To evaluate toxicity of combination therapy (carfilzomib, lenalidomide, and dexamethasone).
* To evaluate disease heterogeneity in relation to clinical outcomes (molecular profiling on bone marrow samples)

Study design:

Randomized multi-center open-label phase 2 trial.

Study population:

Patients with high-risk SMM, age 18 years or older

Intervention (if applicable):

Patients will be treated with KRd combination 9 cycles a 28 days (carfilzomib , lenalidomide , dexamethasone) or Rd combination (lenalidomide , dexamethasone ); followed by extended lenalidomide dosing (for 24 cycles a 28 days).

Primary study parameters/outcome of the study:

- Progression-free survival rate, defined as time from study entry to progression or death, whichever comes first;

Secundary study parameters/outcome of the study (if applicable):

* MRD status after induction cycle 4 and 9,
* Progression-free survival-2 (PFS2), defined at time from randomization to progression after second-line treatment or death, whichever comes first;
* Duration of response (DOR), defined as time from response to progression or death, whichever comes first;
* Overall survival (OS), defined as time from study entry to death from any cause. Patients still alive at the date last contact will be censored;
* Correlation of MRD status with PFS, PFS2, DOR and OS;
* Toxicity of combination therapy (carfilzomib, lenalidomide, and dexamethasone). Nature and extent of the burden and risks associated with participation, benefit and group relatedness (if applicable): Given the high rates of progression specific to the high risk SMM populations and low toxicity profile of combination therapy, risk of exposure does not seem to outweigh the clinical benefit that patients may derive from therapy. More importantly, much of patient morbidity in MM is associated with pain from irreversible skeletal related events. This study aims to treat or cure the disease before irreversible bone damage occurs or before aggressive clinical MM occurs.

Discomfort from venipuncture, bone marrow biopsy, and CT scan is minimal and of limited risk

ELIGIBILITY:
Inclusion criteria

* Patients must have histologically or cytologically confirmed Smoldering Multiple Myeloma based on the 2014 International Myeloma Working Group Criteria(20):
* Serum M-protein ≥3.0 g/dl, or urinary monoclonal protein >500 mg per 24 hours, and/or monoclonal bone marrow plasma cells ≥10-60 %
* Absence of CRAB symptoms:
* anemia: Hemoglobin <6.2 mmol/L (10 g/dl) or a hemoglobin value of >1.2 mmol/L (2 g/dL) below the lower limit of normal
* renal failure: serum creatinine > 2.0 mg/dL or creatinine clearance < 40 ml/min
* hypercalcemia: serum calcium >0·25 mmol/L (>1 mg/dL) higher than the upper limit of normal or >2·75 mmol/L (>11 mg/dL)
* Bone lesions: one or more osteolytic lesions on skeletal radiography, CT, or PET-CT
* Absence of myeloma defining events:
* Involved/uninvolved serum free light chain ratio ≥100 with involved free light-chain concentration ≥10 mg/dl
* Presence of 2 or more focal lesions by MRI (2 of which at least 5 mm)
* Clonal bone marrow plasma cell percentage ≥60%
* Patients must have high risk Smoldering Multiple Myeloma based on the Mayo Clinic and/or the PETHEMA criteria:
* 3 factors of Mayo Clinic criteria:
* Bone marrow plasma cells ≥10 %
* Serum M-protein ≥ 3 g/dl
* Serum free light-chain ratio <0.125 or >8
* And/or 2 factors of PETHEMA criteria:
* Of the plasma cell population ≥95% abnormal plasma cells (presence or absence of CD38, CD56, CD19 and/or CD45)
* Immunoparesis, a reduction (below the lower normal limit) in the levels of 1 or 2 of the uninvolved immunoglobulins (Ig)
* Measurable disease defined by any one of the following:
* Serum monoclonal protein ≥ 1.0 g/dl
* Urine monoclonal protein >200 mg/24 hour
* Serum immunoglobulin free light chain >10 mg/dL AND abnormal kappa/lambda ratio (reference 0.26-1.65)
* Age >18 years
* WHO/ECOG performance status <2 (see Appendix C).
* Patients must have normal organ and marrow function as defined below:
* Absolute neutrophil count >1.0 x109 /L
* Platelets ≥75 ×109 /L
* Hemoglobin ≥10 g/dL (>6.2 mmol/l)
* Total bilirubin <1.5 x institutional upper limit of normal
* AST(SGOT)/ALT(SGPT) ≤3.0 × institutional upper limit of normal
* Creatinine Clearance ≥ 50 ml/min. CrCl will be calculated by Cockcroft-Gault method or eGFR (Modified Diet in Renal Disease [MDRD])
* Females of childbearing potential must have a negative serum or urine pregnancy test within 10 - 14 days prior to entry and again within 24 hours of starting lenalidomide treatment; (see 9.1.4)
* Patients must be willing and capable to use adequate contraception during and after the therapy (all men, all pre-menopausal women) (see 9.1.4.); Patients must be able to adhere to the requirements of the Lenalidomide Clinical Trial Pregnancy Prevention Plan;
* Written informed consent
* Patient is capable of giving informed consent

Exclusion criteria

* Patients with symptomatic multiple myeloma (i.e. having myeloma defining events)
* Amyloid Light-chain (AL) amyloidosis
* Patients who are receiving any other investigational agents.
* Concurrent systemic treatment or prior therapy within 4 weeks for SMM (if a patient has received any previous SMM therapy this must be discussed with the Principal Investigator before inclusion in the trial).

Treatment with corticosteroids for other indications is permitted

* Contraindication to any concomitant medication, including antivirals, anticoagulation prophylaxis, tumor lysis prophylaxis, or hydration given prior to therapy
* History of allergic reactions attributed to immunomodulatory agents and proteasome inhibitors.
* Uncontrolled hypertension or diabetes
* Pregnant or lactating females.
* Significant cardiovascular disease with NYHA grade III or IV symptoms, or hypertrophic cardiomegaly, or restrictive cardiomegaly, or myocardial infarction within 3 months prior to enrollment, or unstable angina, or unstable arrhythmia
* Active hepatitis B or C infection
* Known or suspected HIV infection
* Incidence of gastrointestinal disease that would prevent absorption.
* Significant neuropathy ≥Grade 3 or grade 2 with pain within 14 days of enrollment
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection.
* History of other malignancy (apart from basal cell carcinoma of the skin, or in situ cervix carcinoma) except if the patient has been free of symptoms and without active therapy during at least 5 years
* Major surgery within 1 month prior to enrollment
* Pre-existing pulmonary, cardiac or renal impairement that prevents hydration measures as described at paragraph 9.1.4
* Any psychological, familial, sociological and geographical condition potentially hampering compliance with the study protocol and follow-up schedule.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2018-11-19 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival rate | Until 5 years after randomization or death, whatever comes first
  Time from study entry to progression or death, whichever comes first

SECONDARY OUTCOMES:
MRD status | 9 months
  MRD assessment by immunophenotyping in bone marrow after induction cycles 4 and 9
Progression-free survival-2 (PFS2), | Until 5 years after randomization or death, whatever comes first
  Time from randomization to progression after second-line treatment or death, whichever comes first
Duration of response (DOR), | Until 5 years after randomization or death, whatever comes first
  Time from response to progression or death, whichever comes first
Overall survival (OS) | Until 5 years after randomization or death, whatever comes first
  Time from study entry to death from any cause. Patients still alive at the date last contact will be censored.
MRD status correlation | Until 5 years after randomization or death, whatever comes first
  Correlation of MRD status with PFS, PFS2, DOR and OS
Toxicity of combination therapy with Carfilzomib. Lenalidomide and Dexamethasone | Through induction treatment and extrended treatment, up to 3 years after randomization
  Measured by tabulation of the incidence of adverse events with CTCAE grade 1 or more, separately for induction treatment and for extended treatment, by randomization arm.

CONTACTS AND LOCATIONS:
Overall Officials: A. Broijl, Principal Investigator — Erasmus MC / HOVON
Locations (16):
- Czechia (2):
  - CZ-Brno-UHBRNO, Brno
  - CZ-Ostrava-Poruba-FNO, Ostrava
- Italy (5):
  - IT-Ancona-UMBERTOA, Ancona
  - IT-Bologna-MALPHIGI, Bologna
  - IT-Brescia-SPEDALICIVILI, Brescia
  - IT-Roma-SAPIENZA, Roma
  - IT-Torino-MOLINETTE, Torino
- Netherlands (8):
  - NL-Den Bosch-JBZ, 's-Hertogenbosch
  - NL-Amsterdam-VUMC, Amsterdam
  - NL-Hoofddorp-SPAARNEGASTHUIS, Hoofddorp
  - NL-Leeuwarden-MCL, Leeuwarden
  - NL-Nijmegen-RADBOUDUMC, Nijmegen
  - NL-Rotterdam-ERASMUSMC, Rotterdam
  - NL-Sittard-Geleen-ZUYDERLAND, Sittard
  - NL-Utrecht-UMCUTRECHT, Utrecht
- NO-Oslo-OSLOUH, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: HOVON website — http://www.hovon.nl